CLINICAL TRIAL: NCT03363724
Title: A Retrospective, Multi-Center, Clinical Validation of HaGuide Software Module Accuracy in Mapping Sub-thalamic Nucleus (STN) Boundaries in Parkinson's Disease Patients Who Underwent Deep Brain Stimulation (DBS) Procedure
Brief Title: Validation of HaGuide Software Module Accuracy in Mapping STN Boundaries in Parkinson's Disease Patients Who Underwent DBS Procedure
Status: Completed | Type: Observational
Sponsor: Alpha Omega Engineering Ltd. (Industry)
Collaborators: University of Colorado, Denver (Other); Hadassah Medical Organization (Other); Swedish Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: AO-001
Record Dates: First submitted 2017-11-19; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Parkinson Disease; Deep Brain Stimulation
Keywords: Parkinson Disease; Deep Brain Stimulation; Microelectrodes recording; HaGuide; Alpha Omega Engineering Ltd.
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HaGuide version 1.0 software module: Patients diagnosed with Parkinson's Disease who underwent implantation of DBS electrode in the STN for the treatment of Parkinson's Disease, using the Neuro-Omega device for navigation and procedure's MER digital recorded data is available.
  Interventions: Other: HaGuide version 1.0 software module

INTERVENTIONS:
Other: HaGuide version 1.0 software module

SUMMARY:
HaGuide version 1.0 (Neuro-Omega Ltd.) is a software module add-on to the FDA cleared Neuro-Omega System (K123796). It was designed to facilitate the use of Neuro-Omega's system by automatically mapping visually the depth of STN landmarks intra-operatively. HaGuide algorithm computes and displays the STN entry and exit, as well as introduces a detection of a distinct DLOR-VMNR boundary. HaGuide visual display is added to the UI and it is supplementing and not replacing the previously cleared standard display (visual and audio) of the system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was diagnosed with Parkinson's disease;
2. Patient underwent implantation of DBS electrode in the STN for the treatment of Parkinson's disease, using the Neuro-Omega device for navigation;
3. Procedure's MER digital recorded data is available;

Exclusion Criteria:

1. DBS performed for any other movement disorder other than Parkinson's Disease including Parkinsonism;
2. The recording has a high intensity of noise that will not allow re-analysis using the HaGuide software, in such cases the HaGuide software indicates that the signal is not valid for analysis;
3. Missing data for primary end-point on the respective patient medical chart;
4. The collected data that is used for the validation is with high step size resolution;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Parkinson's Disease who underwent implantation of DBS electrode in the STN for the treatment of Parkinson's Disease, using the Neuro-Omega device for navigation and procedure's MER digital recorded data is available.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
HaGuide vs. Neurosurgeon measurements | 2 weeks
  Percent agreement between HaGuide software measurements and expert Neurosurgeon/Electrophysiologist measurements

SECONDARY OUTCOMES:
DLOR vs. VMNR | 2 weeks
  Length (mm) of Dorso-Lateral Oscillatory Region (DLOR) vs. Ventro-Medial Non-Oscillatory Region (VMNR);
DLOR Entry/exit | 2 weeks
  Entry/exit from DLOR (depth in mm)
STN Length | 2 weeks
  Length of STN track (mm
DBS implant optimal track Identification | 2 weeks
  Percent agreement in DBS implant optimal track Identification by percent agreement between HaGuide and Neurosurgeon choice of optimal track for DBS implant
Sites/Users comparison | 2 weeks
  Sub-group analysis to determine the variation between sites by percent agreement between HaGuide software measurements and expert Neurosurgeon/Electrophysiologist measurements

CONTACTS AND LOCATIONS:
Overall Officials: John A Thompson, Dr., Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No